CLINICAL TRIAL: NCT06434766
Title: A Multicenter Clinical Study on Transcranial Magnetic Stimulation of the Primary Motor Cortex for PTSD Treatment
Brief Title: Multicenter iTBS Neuromodulation for PTSD Treatment
Acronym: TMCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shanghai Mental Health Center (Other); The Affiliated Kangning Hospital of Ningbo University (Unknown); The First Affiliated Hospital of Anhui Medical University (Other); Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: yan2024-0108
Record Dates: First submitted 2024-05-15; First posted 2024-05-30 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2024-09

CONDITIONS: Posttraumatic Stress Disorder
Keywords: iTBS; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Sham stimulation is used as a parallel control group for iTBS group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators and outcomes assessors are all blind to the group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham stimulation (Sham Comparator): A sham coil with exactly the same appearance of active coil is used to compare with active coil. Stimulation dose and frequency is the same as active stimulation.
  Interventions: Device: sham stimulation
- Active stimulation (Active Comparator): An active coil is used to deliver iTBS. The stimulation dose is 20 sessions (1800 pulses per session; 2 sessions a day, at least 1 hour apart) over the course of 2 weeks (10 days to 14 days, allow at most three breaks and only once of the longest interval of 2 days).
  Interventions: Device: intermittent theta-burst stimulation (iTBS)

INTERVENTIONS:
Device: sham stimulation — sham theta-burst transcranial magnetic stimulation
  Arms: Sham stimulation
Device: intermittent theta-burst stimulation (iTBS) — intermittent theta-burst transcranial magnetic stimulation
  Arms: Active stimulation

SUMMARY:
The proposed study aims to evaluate the efficacy of intermittent theta-burst transcranial magnetic stimulation (iTBS) targeting primary motor cortex (M1) as adjunct treatment for PTSD patients. The primary outcome measure includes changes in PTSD symptom severity, with secondary outcome measures focusing on negative moods improvements, quality of life and social/occupation functioning and functional connectivity of the brain.

DETAILED DESCRIPTION:
The proposed study aims to evaluate the efficacy of intermittent theta-burst transcranial magnetic stimulation (iTBS) targeting primary motor cortex as adjunct treatment for PTSD patients.

Compared to traditional repetitive transcranial magnetic stimulation (rTMS), iTBS strategy usually delivers large amounts of pulses in a shorter time period, and its equal efficiency has been demonstrated in several psychiatric disorders such as major depressive disorder (MDD). Through this adequately randomized and sham-controlled study of iTBS for PTSD, this work will provide an alternative and potentially more potent stimulation target for clinical PTSD treatment. This study will also provide a comprehensive assessment of this treatment strategy towards improvements in symptoms, quality of life and brain functioning in PTSD.

The ultimate goal of this study is to develop a non-invasive brain stimulation approach targeting a novel site for alleviating symptoms and improving life quality for PTSD patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 to 65 years old
* Right handedness
* Have a diagnosis of PTSD meeting DSM-5 criteria
* CAPS-5 score>35
* Under stable medication for at least four weeks
* Capable of independently reading and understanding study materials and providing informed consent.

Exclusion Criteria:

* Current (or past if appropriate) significant neurological or medical disorder, or lifetime history of 1) seizure disorder; 2) primary or secondary CNS tumors; 3) stroke; or 4) cerebral aneurysm.
* Primary psychotic disorder, bipolar I disorder, major depressive disorder, or personality disorders
* Lifetime history of attempted suicide or HAMD-17 suicide item (item 3) ≥ 3 points
* Implanted device (deep brain stimulation) or metal in the brain; a pacemaker, extensive dental work, or any magnetic metal implants and upper body tattoos if choose to do fMRI
* Previous experience of rTMS
* Pregnancy/lactation, or planning to become pregnant during the study
* Current under psychological or other physical treatments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD Symptom Severity | Baseline and 4 weeks after finishing treatment
  Change in PTSD symptom severity measured by the Clinician Administered PTSD Scale for DSM-5 (CAPS-5).
  The CAPS-5 is a structured interview designed to make a categorical PTSD diagnosis, as well as to provide a measure of PTSD symptom severity. The structure corresponds to the DSM-5 criteria, with B, C, D and E symptoms rated for both frequency and intensity which are summed to provide severity ratings. Items rated '0' means 'absent' and item rated '4' means 'extreme/incapacitating'. Higher scores indicate more severe PTSD symptoms.

SECONDARY OUTCOMES:
Change in PTSD Symptom Severity | Baseline, 10 times treatment, 20 times treatment, 2 weeks after finishing treatment and 8 weeks after finishing treatment
  Change in PTSD symptom severity measured by the Clinician Administered PTSD Scale for DSM-5 (CAPS-5).
Change in Post-traumatic Stress Disorder Checklist for DSM-5 (PCL-5) Total Score | Baseline, 10 times treatment, 20 times treatment, 2, 4 and 8 weeks after finishing treatment
  The PCL-5 is a 20-item self-report checklist of PTSD symptoms based closely on the DSM-5 criteria. Respondents rate each item from 0 ("not at all") to 4 ("extremely") to indicate the degree to which they have been bothered by that particular symptom over the past month (or past week if using the PCL-5 weekly). A total symptom severity score (range: 0-80) can be obtained by summing the scores for each of the 20 items, with higher scores indicating more severe PTSD symptoms.
Change in The Quick Inventory of Depressive Symptomatology Self Report (QIDS-SR) Score | Baseline, 10 times treatment, 20 times treatment, 2, 4 and 8 weeks after finishing treatment
  The IDS-SR is a 30-item questionnaire measuring depressive symptoms. Each item has four statements that reflect various degrees of symptom severity, scored on a four-point scale from 0 to 3. The 16-item Quick Inventory of Depressive Symptomatology (QIDS) is a new measure of depressive symptom severity derived from the 30-item IDS-SR and has highly acceptable psychometric properties.
Change in The Personal Social Performance (PSP) scale | Baseline, 10 times treatment, 20 times treatment, 2, 4 and 8 weeks after finishing treatment
  The Personal and Social Performance Scale (PSP) is a 100-point single-item rating scale that assesses four important domains of patients with mental disorders. The four main areas include (a) socially useful activities, including work and study; (b) personal and social relationships; (c) self-care; and (d) disturbing and aggressive behaviors.
change in Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) | Baseline, 10 times treatment, 20 times treatment, 2, 4 and 8 weeks after finishing treatment
  Q-LES-Q-SF is a patient-reported 16-item instrument that measures the degree of enjoyment and satisfaction in daily life over the past week. Individual items are rated on a scale from 1-5 ('very poor', 'poor', 'fair', 'good', or 'very good'). The Q-LES-Q-SF total score is the sum of the first 14 item scores (i.e. excluding medication satisfaction and overall life satisfaction and contentment) with a higher score indicating greater satisfaction (range = 14-70).
Change in neural activity pattern and functional connectivity of the brain based on fMRI | Baseline, 20 times treatment, 4 weeks after finishing treatment
  Structural, resting-state and task-based fMRI will be performed if the participant agree. During task-fMRI, the participant will listen to a script around one minute recorded during his/her first interview, describing the traumatic experience in details. The participant will be instructed to recall the traumatic experience vividly during the task-fMRI. Brain activity patterns and connectivity network will be presented and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shen, M.D., Ph.D., Principal Investigator — Shanghai Mental Health Center; Chang Yu, M.D., Principal Investigator — The Affiliated Kangning Hospital of Ningbo University; Kai Wang, M.D., Ph.D., Principal Investigator — The First Affiliated Hospital of Anhui Medical University; Xiaoming Li, M.D., Ph.D., Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (5):
- China (5):
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Anhui Medical University, Hangzhou, Zhejiang
  - Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Affiliated Kangning Hospital of Ningbo University, Ningbo, Zhejiang
  - Tongji Hospital of Tongji University, Shanghai

IPD SHARING:
Plan to Share IPD: No